CLINICAL TRIAL: NCT00094536
Title: A Study to Evaluate the Effectiveness of Extended Treatment Regimens With the Her Option® Cryoablation Therapy System for Treatment of Menorrhagia
Brief Title: Evaluation of Modified Treatment Regimens for Treatment of Heavy Menstrual Bleeding Using the HerOption® System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CooperSurgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AMS043
Record Dates: First submitted 2004-10-20; First posted 2004-10-21 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; Excessive Uterine Bleeding; Cryoablation; Menstrual disorder; Endometrial ablation; Abnormal uterine bleeding; Dysfunctional uterine bleeding
MeSH Terms: conditions — Menorrhagia; Menstruation Disturbances; Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Extended Treatment Regimen (Experimental): Extended treatment regimens using the Her Option Endometrial Cryotherapy System to more effectively ablate the endometrial lining, reducing menstrual levels to normal or less.
  Interventions: Device: Extended treatment regimen using Her Option Cryotherapy

INTERVENTIONS:
Device: Extended treatment regimen using Her Option Cryotherapy — Extended treatment regimens using the Her Option Endometrial Cryotherapy System to more effectively ablate the endometrial lining, reducing menstrual levels to normal or less.
  Other Names: Her Option

SUMMARY:
The Her Option® Cryoablation Therapy System is a closed-loop cryosurgical device that is used to ablate the endometrial lining in pre-menopausal women with menorrhagia (excessive menstrual bleeding) due to benign causes. This is a non-incisional procedure, which can be performed in a physicians office with minimal sedation.

Initial FDA clinical studies were conducted with a two-freeze treatment pattern consisting of a 4 minute freeze with the Cryoprobe positioned in one cornu followed by a second freeze of 6 minutes with the Cryoprobe repositioned in the contralateral cornu.

Since completion of the early studies, many physicians have experimented with varying freeze patterns using longer freeze durations and/or additional freezes at the fundus and the lower uterine segment. The results, as reported in the literature, indicate that these extended freeze patterns produce significantly better results than the original regimen.

DETAILED DESCRIPTION:
American Medical Systems, Inc. (AMS) hypothesized that the original treatment pattern used to support a previous FDA approval for the Her Option® Cryoablation Therapy System for Treatment of abnormal uterine bleeding was not optimal and that extended freeze regimens will result in improved outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal adult women 30 years of age or older who have completed childbearing
* Heavy or prolonged menstrual bleeding
* Willing and able to complete all follow-up exams as required by protocol

Exclusion Criteria:

* Known or suspected endometrial cancer or pre-malignant change of the endometrium
* Untreated cervical dysplasia
* Hereditary malformations of the uterine cavity that would prevent insertion and/or placement of the cryoprobe
* Uterine myomas > or = to 3 cm in diameter
* Past history of invasive treatment for abnormal uterine bleeding or uterine myomas
* History of classical (not low transverse incision) cesarean section
* Active genital or urinary tract infection or acute pelvic inflammatory disease (PID)
* Intrauterine device (IUD) in place
* Other medical conditions could be exclusionary upon evaluation for study treatment

Ages: 30 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Kelly Roy, M.D., P.C., Phoenix, Arizona
  - Institute for Women's Health & Body, Wellington, Florida
  - Lahey Clinic, Burlington, Massachusetts
  - Valley OB/GYN, Saginaw, Michigan
  - Center for Endometrial Ablation, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Jose Manjon, M.D. (Private practice), Camp Hill, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced 8/13/04, and was completed 1/20/06, with final 3-year follow-up occurring on 3/17/09. Assessments occurred at gynecologic offices. The majority of procedures occurred in the office setting, and the remainder in the ASC setting.
Pre-assignment Details: Subjects were consented and assessed for inclusion/exclusion; qualified subjects underwent treatment and are considered the intent-to-treat group.
  Sample size was targeted for 76 subjects, however FDA granted the request for additional subjects to undergo treatment if consented at the time of completion of enrollment.
Groups:
- Extended Treatment Regimen: Extended treatment regimens using the Her Option Endometrial Cryotherapy System.
Period: Inclusion Exclusion Evaluation
Arm/Group | Extended Treatment Regimen
Started | 106
Completed | 82
Not Completed | 24
Not completed — Did not qualify for study treatment | 24
Period: Treatment and Follow-up
Arm/Group | Extended Treatment Regimen
Started | 82 (82 subjects qualified for and underwent the study treatment.)
12 Month Follow-up | 69 (69 subjects were evaluated at 1-year post-treatment for the primary endpoint of success.)
24 Month Follow-up | 53
36 Month Follow-up | 51
Completed | 51 (51 subjects successfully completed the study.)
Not Completed | 31
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 9
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 1
Not completed — Subject non-compliance | 9
Not completed — Unable to attend visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Extended Treatment Regimen
Number analyzed (Participants) | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 79
  More than one race | 2
  Unknown or Not Reported | 0
  Hispanic or Latino | 9
Region of Enrollment [Number; unit: participants]
  United States | 106

OUTCOME MEASURES:

1. Primary Outcome: Success (Reduction in Menstruation to Normal Levels)
Description: Success is defined as a pictorial bleeding assessment chart (PBAC) score of ≤ 75 at 1-year post-treatment; a score which corresponds to normal menstruation levels.
Time Frame: 1 Year
Population: Intention-to-Treat Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Treatment Regimen
Number analyzed (Participants) | 82
Participants | 59
Statistical Analysis 1: Comparison: Extended Treatment Regimen; Test type: Superiority or Other; p = .271, 1-sided z-test; 1-sided z-test with continuity correction (pooled)

ADVERSE EVENTS:
Time Frame: Adverse events were both passively and actively collected and assessed throughout the study, up to 3-years post-treatment.
Arm/Group | Extended Treatment Regimen
Serious Adverse Events (participants affected / at risk) | 19/82
Other Adverse Events (participants affected / at risk) | 16/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Treatment Regimen (N=82)
Adnexial mass/cyst (Reproductive system and breast disorders) | 1 (1)
Bicep Tendon Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer - Breast (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Failed Steriliztion Device Placement (Surgical and medical procedures) | 1 (1)
Hematometria (Reproductive system and breast disorders) | 1 (1)
Labial Hypertrophy Surgery (Surgical and medical procedures) | 1 (1)
Lumbar Fusion Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Menorrhagia/Lack of Efficacy (Reproductive system and breast disorders) | 6 (6)
Polycystic Ovarian Syndrome (Reproductive system and breast disorders) | 1 (2)
Shoulder Slap Lesion Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Incontinence Surgery (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Uterine Perforation During Sterilization Procedure (Surgical and medical procedures) | 1 (1)
Umbilical Hernia Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Treatment Regimen (N=82)
Pain/Discomfort - Pelvic (Reproductive system and breast disorders) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4)
Vaginal Infection (Reproductive system and breast disorders) | 4 (4)
Endometritis (Reproductive system and breast disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The primary endpoint was assessed using a validated diary completed by the subject prior to each visit, which has inherent weaknesses as an objective measure of blood loss.

Use of historical control limits comparison of outcomes across studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No